CLINICAL TRIAL: NCT05652868
Title: A Phase 1 Multicenter Dose Escalation and Dose Expansion Study of Antibody-Drug Conjugate MYTX-011 in Subjects With Non-Small Cell Lung Cancer - KisMET-01
Brief Title: Clinical Study of Antibody-Drug Conjugate MYTX-011 in Subjects With Non-Small Cell Lung Cancer
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Business decision
Sponsor: Mythic Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: MYTX-011-01; KisMET-01 (Other: Mythic Therapeutics)
Record Dates: First submitted 2022-11-29; First posted 2022-12-15 (Actual); Last update posted 2025-12-16 (Actual); Status verified 2025-11

CONDITIONS: NSCLC; NSCLC Stage IV; NSCLC Stage IIIB; Non-Small Cell Lung Cancer; Advanced Non-Small Cell Squamous Lung Cancer; Advanced Non-Small Cell Lung Cancer; Advanced Non-Small Cell Non-Squamous Lung Cancer
Keywords: cMET; MYTX-011; Mythic; MET; MYTX011; ADC; KisMET-01
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (9):
- Part 1 Dose Escalation (Experimental): Part 1 patients will receive MYTX-011.
  Interventions: Drug: MYTX-011
- Part 2 Cohort A (Experimental): Part 2 Cohort A patients will be randomized to two different dose levels of MYTX-011. Doses to be determined after completion of Part 1.
  Interventions: Drug: MYTX-011
- Part 2 Cohort B (Experimental): Part 2 Cohort B patients will receive MYTX-011 at the recommended phase 2 dose.
  Interventions: Drug: MYTX-011
- Part 2 Cohort C (Experimental): Part 2 Cohort C patients will receive MYTX-011 at the recommended phase 2 dose.
  Interventions: Drug: MYTX-011
- Part 2 Cohort D (Experimental): Part 2 Cohort D patients will receive MYTX-011 at the recommended phase 2 dose.
  Interventions: Drug: MYTX-011
- Part 2 Cohort E (Experimental): Part 2 Cohort E patients will receive MYTX-011 at the recommended phase 2 dose.
  Interventions: Drug: MYTX-011
- Part 2 Cohort B2 (Experimental): Part 2 Cohort B2 patients will be randomized to two different dose levels of MYTX-011. Doses to be determined after completion of Part 1
  Interventions: Drug: MYTX-011
- Part 2 Cohort E2 (Experimental): Part 2 Cohort E2 patients will be randomized to two different dose levels of MYTX-011. Doses to be determined after completion of Part 1
  Interventions: Drug: MYTX-011
- Part 2 Cohort F (Experimental): Part 2 Cohort F patients will receive MYTX-011 at the recommended phase 2 dose.
  Interventions: Drug: MYTX-011

INTERVENTIONS:
Drug: MYTX-011 — MYTX-011 will be administered as an intravenous infusion every 21 days.

SUMMARY:
This is a Phase I open label multi-center study to evaluate the safety, tolerability, pharmacokinetics and preliminary effectiveness of the investigational drug MYTX-011 in patients with locally advanced, recurrent or metastatic NSCLC. MYTX-011 is in a class of medications called antibody drug conjugates (ADCs). MYTX-011 is composed of a pH-dependent anti-cMET antibody and the potent antimicrotubule drug monomethyl auristatin E (MMAE).

DETAILED DESCRIPTION:
The study will be conducted in 2 parts. Part 1 will assess the safety and tolerability of MYTX-011 and identify the dose to be studied in Part 2. Part 2 will include subjects with NSCLC with cMET overexpression or MET amplification/exon 14 skipping mutations, populations with a current unmet medical need.

ELIGIBILITY:
Inclusion Criteria:

Part 1:

* Histologically or cytologically confirmed locally advanced, recurrent or metastatic NSCLC and have received available standard of care therapy.
* There is no limit on the number of prior therapies that can have been received.

Part 2 Cohorts A-D and F

1. Known to not have an actionable EGFR mutation. Subjects with or without other driver mutations are permitted to enroll.
2. Must have received (or be ineligible for) available standard of care therapy.
3. Must have progressed on at least 1 line of prior systemic therapy in the locally advanced/metastatic setting. Note: multiple TKIs for the same actionable mutation count as 1 line of therapy. Rechallenge of the same therapy regimen within 6 months of discontinuation date of the therapy is not considered a separate line of therapy. Maintenance therapy is not considered a separate line of therapy. Adjuvant and neoadjuvant therapies count as 1 line of therapy if given within 6 months before study entry. The same rules above apply to all inclusion/exclusion criteria regarding prior lines of therapy.
4. Subjects without any actionable gene alteration: must have progressed on (or be considered ineligible for), or be intolerant to, platinum-based chemotherapy and immune checkpoint inhibitor (as monotherapy or in combination with chemotherapy) and have not received more than 2 lines of prior systemic therapy in the locally advanced/metastatic setting.
5. Subjects with actionable gene alterations (other than EGFR) for which immune checkpoint inhibitor therapy is not standard of care (e.g., anaplastic lymphoma kinase [ALK] translocation): must have progressed on (or be considered ineligible for), or be intolerant to, anticancer therapy targeting driver gene alterations and platinum-based chemotherapy and have not received more than 3 lines of prior systemic therapy in the locally advanced/metastatic setting.
6. Subjects with actionable gene alterations (other than MET exon 14 skipping mutation) for which immune checkpoint inhibitor is standard of care: must have progressed on (or be considered ineligible for), or be intolerant to, anticancer therapy targeting driver gene alteration and platinum-based chemotherapy, and also progressed on (or be considered ineligible for) or be intolerant to immune checkpoint inhibitor(as monotherapy or in combination with platinum-based chemotherapy, and have not received more than 3 lines of prior systemic therapy in the locally advanced/metastatic setting.
7. Subjects with MET exon 14 skipping mutation must have progressed on, or be intolerant to, at least one MET TKI if available, and have not received more than 2 lines of prior systemic therapy in the locally advanced/metastatic setting.

Part 2:

Cohort A:

* Have histologically or cytologically confirmed locally advanced, recurrent (and not a candidate for curative therapy), or metastatic non-squamous NSCLC without EGFR mutation.
* Tumor sample with high cMET expression by IHC confirmed by central laboratory testing.

Cohort B:

* Have histologically or cytologically confirmed locally advanced, recurrent (and not a candidate for curative therapy), or metastatic non-squamous NSCLC without EGFR mutation.
* Tumor sample with intermediate cMET expression by IHC confirmed by central laboratory testing.

Cohort B2

* Have histologically or cytologically confirmed locally advanced, recurrent (and not a candidate for curative therapy), or metastatic non-squamous NSCLC without EGFR mutation.
* Tumor sample with intermediate cMET expression by IHC confirmed by central laboratory testing.

Cohort C:

* Have histologically or cytologically confirmed locally advanced, recurrent (and not a candidate for curative therapy), or metastatic squamous NSCLC without EGFR mutation.
* Tumor sample with cMET expression by IHC confirmed by central laboratory testing.

Cohort D:

* Have histologically or cytologically confirmed locally advanced, recurrent (and not a candidate for curative therapy), or metastatic non-squamous or adenosquamous NSCLC without EGFR mutation.
* Tumor sample with low cMET expression on tumor biopsy confirmed centrally by IHC that does not meet inclusion criteria for Cohorts A, B, or B2.

Cohort E:

* Have histologically or cytologically confirmed locally advanced, recurrent (and not a candidate for a curative therapy), or metastatic NSCLC with actionable EGFR mutations.
* Tumor sample with high or intermediate cMET expression by IHC confirmed by central laboratory testing.
* Must have received an available standard of care therapy and have progressed on at least 1 and no more than 3 lines of prior systemic therapy in the locally advanced/metastatic setting.

Cohort E2

* Have histologically or cytologically confirmed locally advanced, recurrent (and not a candidate for curative therapy), or metastatic NSCLC with actionable EGFR mutations.
* Tumor sample with high or intermediate cMET expression by IHC confirmed by central laboratory testing.
* Must have received an available standard of care therapy and have progressed on at least 1 line and no more than 3 lines of prior systemic therapy in the locally advanced/metastatic setting.

Cohort F

* Have histologically or cytologically confirmed locally advanced non-squamous or adenosquamous NSCLC without EGFR mutation.
* Have ultra-low cMET expression on tumor biopsy confirmed centrally by IHC that does not meet inclusion criteria for Cohorts A,B, B2, or D.

All patients (Part 1 and Part 2)

Inclusion Criteria:

* Patient has at least one measurable lesion per RECIST 1.1
* ECOG performance status 0 or 1
* For women of childbearing potential and men with partners of childbearing potential, agreement to use a highly effective method of birth control for the duration of the study treatment and for at least 6 months after the last dose of study drug.
* Able to provide informed consent, and willing and able to comply with study protocol requirements

Exclusion Criteria:

Radiation to the lung within 6 weeks prior to screening. For all other sites (except lung), therapeutic or palliative radiation within 2 weeks prior to the first dose of study drug. Must have recovered from all radiation-related toxicity.

Major surgery within 28 days of first dose of study drug administration.

Untreated, uncontrolled central nervous system (CNS) metastases and/or leptomeningeal disease.

* History of interstitial lung disease or pneumonitis that required treatment with systemic steroids or evidence of active interstitial lung disease or pneumonitis. A history of prior radiation pneumonitis in the radiation field (fibrosis) is permitted.
* Clinically significant systemic illness that could pose undue risk to the subject or confound the ability to interpret study results.
* Active infection requiring IV antibiotics, antivirals, or antifungal medication within 14 Days of Cycle 1 Day 1
* Neuropathy > Grade 1
* History of cirrhosis, hepatic fibrosis, esophageal or gastric varices, or other clinically significant liver disease.
* Active or chronic corneal disorder
* Conditions that may interfere with assessment of vision, such as monocular status or severe visual impairment in 1 or both eyes

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 227 (Actual)
Dates: Start 2023-03-23 (Actual); Primary Completion 2025-10-31 (Actual); Study Completion 2025-11-07 (Actual)

PRIMARY OUTCOMES:
Part 1: Number of patients with dose limiting toxicity (DLT) | Up to Day 21
  The dose limiting toxicities will be based on number and severity of treatment-related adverse events.
Part 2: Number of patients with tumor response | 2 years
  The overall response rate will be based on number of complete responses and partial responses.

SECONDARY OUTCOMES:
Part 1: Pharmacokinetic (PK) parameter (Total ADC) | 24 months
  Total ADC
Part 1: Pharmacokinetic (PK) parameter (Total antibody) | 24 months
  Total antibody
Part 1: Pharmacokinetic (PK) parameter (Free MMAE) | 24 months
  Free MMAE
Part 1: ADA | 24 months
  Presence of anti-drug antibodies
Part 1: ORR | 24 months
  Complete response + partial response
Part 1: DOR, TTR, DCR | 2 years
  Duration of response in patients that achieve CR or PR, time to response, best overall response and disease control rate
Part 1: PFS | for up to 2 years after end of treatment
  Progression free survival
Part 1: OS | for up to 2 years after end of treatment
  Overall survival

CONTACTS AND LOCATIONS:
Overall Officials: Ting Wu, MD MSc, Study Director — Mythic Therapeutics
Locations (55):
- United States (17):
  - University of California San Diego, La Jolla, California
  - UCLA, Los Angeles, California
  - Hoag Memorial Hospital Presbyterian, Newport Beach, California
  - Piedmont Physicians Medical Oncology, Atlanta, Georgia
  - Winship Cancer Institute, Emory University, Atlanta, Georgia
  - Massachusetts General Hospital, Boston, Massachusetts
  - Washington University School of Medicine in St. Louis, St Louis, Missouri
  - Nebraska Cancer Specialists, Omaha, Nebraska
  - Atlantic Health System, Morristown, New Jersey
  - NYU Langone Medical Center, New York, New York
  - UPMC Hillman Cancer Center, Pittsburgh, Pennsylvania
  - MUSC Hollings Cancer Center, Charleston, South Carolina
  - Sarah Cannon Research Institute, Nashville, Tennessee
  - MD Anderson Cancer Center, Houston, Texas
  - NEXT Oncology, Fairfax, Virginia
  - Fred Hutchinson Cancer Center, Seattle, Washington
  - Medical College of Wisconsin, Milwaukee, Wisconsin
- Australia (4):
  - Blacktown Hospital, Blacktown, New South Wales
  - Chris O'Brien Lifehouse, Camperdown, New South Wales
  - Queen Elizabeth Hospital, Adelaide, South Australia
  - Cancer Research SA, Adelaide, South Australia
- France (7):
  - Institut Bergonié-Bordeaux, Bordeaux
  - Centre Léon Bérard - Lyon, Lyon
  - APHM - Hopital de la Timone, Marseille
  - Institut de Cancérologie de l'Ouest (ICO institute)-St Herblain, Nantes
  - INSTITUT Curie (lead), Paris
  - Oncopole Claudius Regaud, IUCT-Oncopole, Toulouse
  - Gustave Roussy Institute, Villejuif
- South Korea (8):
  - Seoul National University Hospital, Seoul, MA
  - Kosin Univ. Gospel Hospital, Busan
  - Chungbuk National Univ. Hospital, Incheon
  - Gachon University, Seongnam
  - National Cancer Center, Seoul
  - Samsung Medical Center, Seoul
  - Severance Hospital, Seoul
  - St. Vincent Hospital, Suwon
- Spain (9):
  - Instituto Oncológico Dr Rosell (IOR) - Hospital Univ. Dexeus, Barcelona
  - START Barcelona-HM CIOCC Early Phase Program, Barcelona
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Universitario Ramón y Cajal, Madrid
  - START Centro Integral Oncologico Calra Campal, Madrid
  - START Madrid-FJD, Hospital Fundación Jiménez Díaz, Madrid
  - Hospital Quirónsalud Málaga, Málaga
  - Hospital Clinico Universitario de Valencia, Valencia
  - Hospital Universitario Lozano Blesa, Zaragoza
- Taiwan (6):
  - Taichung Veterans General Hospital, Taichung, MA
  - National Cheng Kung University Hospital, Tainan
  - National Taiwan University Hospital, Taipei
  - Taipei Medical University Hospital, Taipei
  - National Taiwan University Cancer Centre, Taipei
  - National Taiwan University Hospital Hsin-Chu Branch, Zhubei
- United Kingdom (4):
  - Beatson West of Scotland Cancer Centre, Glasgow
  - University College London Hospitals NHS Foundation Trust, London
  - Newcastle upon Tyne Hospital (NHS), Newcastle
  - Churchill Hospital - Oxford University Hospitals, Oxford

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: CSR
Time Frame: At the conclusion of the study

REFERENCES:
- [Derived] Gera N, Fitzgerald KM, Ramesh V, Patel P, Kanojia D, Colombo F, Kien L, Aoyama S, Xu L, Jean J, Deshpande AM, Comb WC, Chittenden T, Fiske BP. MYTX-011: A pH-Dependent Anti-c-MET Antibody-Drug Conjugate Designed for Enhanced Payload Delivery to c-MET-Expressing Tumor Cells. Mol Cancer Ther. 2024 Sep 4;23(9):1282-1293. doi: 10.1158/1535-7163.MCT-23-0784. PMID 38684230

DOCUMENTS (2):
  • Study Protocol (2025-08-29): https://cdn.clinicaltrials.gov/large-docs/68/NCT05652868/Prot_000.pdf
  • Statistical Analysis Plan (2025-05-15): https://cdn.clinicaltrials.gov/large-docs/68/NCT05652868/SAP_001.pdf